CLINICAL TRIAL: NCT04651374
Title: COVID-19 And Geko Evaluation: The CAGE Study
Acronym: CAGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study site was unable to proceed with recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISS-COV-002
Record Dates: First submitted 2020-11-27; First posted 2020-12-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Covid19
Keywords: ICU; Covid 19; C19; Coronavirus; geko; Deep venous thrombosis; DVT
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial of 20 participants in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geko Device (Experimental): Confirmed Covid-19 positive patients will be randomized to either applying the Geko device arm or the no device arm.
  Interventions: Device: geko T3
- No Device (No Intervention): Confirmed Covid-19 positive patients will be randomized to either applying the Geko device arm or the no device arm.

INTERVENTIONS:
Device: geko T3 — The device stimulates the peroneal nerve.It will be applied for the entire duration of ICU stay and replaced once every 24 hours.
  Other Names: NMES
  Arms: Geko Device

SUMMARY:
The primary objectives of this pilot study protocol are to assess safety and feasibility of using the geko™ device in COVID-19.

Regarding safety to patients, we will measure the rate of adverse events, primarily local site irritation or discomfort. Feasibility will be measured on the basis of recruitment; ability to enroll sufficient number of patients meeting criteria. Protocol adherence will be observed as the ability to deliver the study intervention to the patients randomized to the treatment arm within the prescribed timeline and ability to complete the course of treatment. Additionally, we plan to measure patient outcomes such as ICU admission and death. The findings of this study have the potential to decrease the complications seen in COVID-19 infections.

DETAILED DESCRIPTION:
On March 11, 2020, a global pandemic was declared by the World Health Organization. A novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was identified as the cause of the COVID-19 pandemic. SARS-CoV-2 infection has quickly become one of the fastest growing and deadliest diseases to surface due to its high death rate and ability to replicate and spread readily from people without symptoms. Recent evidence indicates that critically ill patients with COVID-19 experience a high risk of blood clots. Deep leg vein blood clots can travel to the lungs and cause severe lung failure and death. The geko™ device is a simple device that increases the return of blood flow from the lower legs and potentially decrease the risk of lung blood clots. Investigators believe the geko™ device may have an important benefit in COVID-19 patients by decreasing the risk of lung clots and decrease the risk of respiratory failure which is often the cause of death in COVID-19 patients. In this study, Investigators plan to study the effect of using the geko™ device in COVID-19 patients and measure patient outcomes such as ICU admission and death. The findings of this study have the potential to decrease the complications seen in COVID-19 infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients who test positive for Covid-19

Exclusion Criteria:

* Patients who are unlikely to be adherent or cannot tolerate the therapy (self-report)
* Prior above or below knee amputation
* A history of prior Deep Venous Thrombosis (DVT) or Venous Thromboembolism (VTE),
* Those patients being treated with full dose therapeutic anticoagulation.
* Patients with pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | Within a two year period
  Feasibility will be measured on the basis of recruitment; ability to enroll sufficient number of patients meeting criteria
Safety of device: AE | From ICU admission to discharge or death in ICU up to 28 days whichever comes first.
  We will measure the rate of adverse events, primarily local site irritation or discomfort
Protocol Adherence | From ICU admission to discharge or death in ICU up to 28 days whichever comes first.
  We will assess our ability to deliver the study intervention to the patients randomized to the treatment arm within the prescribed timeline and ability to complete the course of treatment

SECONDARY OUTCOMES:
Mortality | From date of admission to discharge from ICU or death in hospital assessed up to a 28 days whichever comes first.
  The impact of the geko™ device on patient outcomes in critically ill COVID-19 patients.
Morbidity | From date of admission to discharge from ICU assessed up to a 28 days whichever comes first.
  The impact of the geko™ device on patient outcomes in critically ill COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Mele, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No